CLINICAL TRIAL: NCT02772510
Title: Upper Extremity Rehabilitation Using Game-based Virtual Reality Rehabilitation System (Smart Glove System) With Functional Electrical Stimulation for Stroke Patients : Randomized Controlled Trial
Brief Title: Upper Extremity Rehabilitation Using Game Rehabilitation System With Functional Electrical Stimulation for Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Manager, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRC-2015-01-004
Record Dates: First submitted 2016-05-08; First posted 2016-05-13 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; Hand; Game; Functional electrical stimulation; Virtual reality
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smart glove system with functional electrical stimulation (Experimental): game-based virtual reality rehabilitation combined with functional electrical stimulation for upper extremity
  Interventions: Device: Smart glove system with functional electrical stimulation
- Functional electrical stimulation (Active Comparator): functional electrical stimulation on upper extremity
  Interventions: Device: Functional electrical stimulation

INTERVENTIONS:
Device: Smart glove system with functional electrical stimulation — Game-based virtual reality rehabilitation system (Smart glove system) combined with functional electrical stimulation on distal upper extremity
  Arms: Smart glove system with functional electrical stimulation
Device: Functional electrical stimulation — Functional electrical stimulation on distal upper extremity
  Arms: Functional electrical stimulation

SUMMARY:
The purpose of the present study was to investigate the effects of game-based virtual reality rehabilitation combined with functional electrical stimulation on distal upper extremity function, and compare the findings to those of functional electrical stimulation in stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* first-ever ischemic or hemorrhagic stroke
* wrist extensor of medical research council scale 1~3
* No clinical evidence of limited passive range of motion of affected wrist

Exclusion Criteria:

* age <18 years
* severe aphasia resulting in communication difficulties confounding intervention and outcome measures
* severe cognitive impairment resulting cooperation difficulties
* spasticity > modified Ashworth scale 1+

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Wolf Motor Function Test | 4 weeks from baseline
Fugl-Meyer Assessment-hand & wrist | 4 weeks from baseline

SECONDARY OUTCOMES:
Wolf Motor Function Test | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
Box and Block Test | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  number of block transferred by hand from one box to other box.
Fugl-Meyer Assessment upper extremity | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  global assessment of upper extremity impairment
Stroke Impact Scale | baseline, 4 weeks after baseline
Motor Activity Log | baseline, 4 weeks after baseline
Medical research council scale of elbow flexion/extension | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
Medical research council scale of wrist flexion/extension | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
Range Of Motion of elbow flexion/extension | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
Range Of Motion of wrist flexion/extension | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
Brunnstrom stage | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  It represent the recovery status among stroke patients
Jebsen-Taylor hand function test | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
Modified Ashworth scale of elbow flexor/extension | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
Modified Ashworth scale of wrist flexion/extension | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
Modified Tardieu scale of elbow flexor/extension | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
Modified Tardieu scale of wrist flexion/extension | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
Adverse events | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, MS, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SH, Lee JY, Kim MY, Jeon YJ, Kim S, Shin JH. Virtual Reality Rehabilitation With Functional Electrical Stimulation Improves Upper Extremity Function in Patients With Chronic Stroke: A Pilot Randomized Controlled Study. Arch Phys Med Rehabil. 2018 Aug;99(8):1447-1453.e1. doi: 10.1016/j.apmr.2018.01.030. Epub 2018 Mar 2. PMID 29505744